CLINICAL TRIAL: NCT06115759
Title: A Randomized Clinical Trial to Study the "T-REX Twente Regimen" (Thoracic Surgery Rehabilitation Experts Twente) on Quality of Life and Mobilisation Activities for Cardiac Surgery Patients After Median Sternotomy, Compared to Usual Care
Brief Title: RCT on T-REX Twente Regimen Effects on Quality of Life and Mobilisation for Cardiac Surgery Patients After Sternotomy
Acronym: T-REX Twente
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Spectrum Twente (Other)
Collaborators: Foothills Medical Centre (Other)
Responsible Party: Principal Investigator, Frank Halfwerk, Assistant Professor and Technical Medical Doctor in Cardio-Thoracic Surgery, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T-REX Twente; CCMO-ABR 78107 (Other: CCMO); 56700 (Other: CCMO Research with human participants - Overview of medical research in the Netherlands (https://onderzoekmetmensen.nl))
Record Dates: First submitted 2023-10-18; First posted 2023-11-03 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Sternotomy; Cardiovascular Diseases; Physical Inactivity; Quality of Life; Surgery
Keywords: Sternotomy; Cardiac Surgical Procedures; Cardiac Rehabilitation; Early Ambulation
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be actively informed on their study arm, but will receive conventional or interventional rehabilitation instructions, and might be able to deduct their allocation arm.
  The researcher will be blinded for intervention or control group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-REX Twente (Experimental): The intervention group receives the new T-REX Twente precautions, allowing for more independent activities through the use of the tube model (keeping elbows close to the sides).
  Interventions: Behavioral: T-REX Twente precautions
- Usual care (Active Comparator): The control group is not allowed to lift, push, or pull for the first 6 weeks. There is little to no evidence for the current strict precautions currently implemented in the department.
  Interventions: Behavioral: Usual (restrictive) sternal precautions

INTERVENTIONS:
Behavioral: T-REX Twente precautions — The intervention group receives the new T-REX Twente precautions, allowing for more independent activities through the use of the tube model (keeping elbows close to the sides).
  Other Names: The T-REX Twente precautions are inspired on the Keep Your Move in the Tube (KYMITT) principle, and adjusted and improved to our local setting
  Arms: T-REX Twente
Behavioral: Usual (restrictive) sternal precautions — The control group is not allowed to lift, push, or pull for the first 6 weeks. There is little to no evidence for the current strict precautions currently implemented in the department.
  Arms: Usual care

SUMMARY:
The goal of this study is whether the T-REX Twente precautions have a positive impact on the quality of life (MAcNew QLMI), level of physical activity, and reduction of fear of movement in heart patients after a total median sternotomy compared to the (current) standard precautions? Do these precautions also have no adverse effects on pain, wound healing, and/or postoperative complications?

Participants will be instructed by the physiotherapist to both groups immediately postoperatively and are constantly repeated by the involved disciplines during the hospital stay.

The control group is not allowed to lift, push, or pull for the first 6 weeks. There is little to no evidence for the current strict precautions currently implemented in the department.

The intervention group receives the new T-REX Twente precautions, allowing for more independent activities through the use of the tube model (keeping elbows close to the sides).

All patients receive three questionnaires (MacNew QLMI, Numeric Pain Rating Scale, and Tampa Scale for Kinesiophobia) preoperatively, on the 4th day postoperatively, on the first day of cardiac rehabilitation, and at the end of cardiac rehabilitation, taking approximately 10 minutes each time. Additionally, during the clinical admission immediately postoperatively, two AX3 accelerometers are placed on the patient, one lateroproximal on the right upper arm and one anterodistal on the right upper leg.

Researchers will compare heart patients after a total median sternotomy with T-REX Twente precautions (intervention group) to the (current) standard precautions (control group).

DETAILED DESCRIPTION:
Each year, more than 1000 open-heart surgeries (OHO) are performed at Thorax Centrum Twente (TCT), with 860 of them involving a total median sternotomy. Some patients present themselves at the cardiac care unit with unexplained complaints after discharge, possibly caused by anxiety and insecurity.

There is no consensus regarding postoperative sternal precautions following a total median sternotomy. Studies in the United States and Canada have indicated that these precautions might be too strict, and alternative, less restrictive precautions through the use of the "Keep your Move in the Tube" (KYMITT) approach have been shown safe and without adverse consequences.

Although no statistically significant differences were observed in all outcomes, patients following the new approach (KYMITT) reported fewer issues with functional mobility.

This is a prospective randomized double blind study, collecting data from patients undergoing a total median sternotomy from November 2023 to November 2025 at TCT and concurrently participating in outpatient cardiac rehabilitation under the guidance of TCT.

Previous research using the MacNew quality of life questionnaire among 677 cardiac rehabilitation patients indicated that the difference in response was normally distributed with a standard deviation of 0.25. The KvL-H is the Dutch (validated) translation of the MacNew QLMI. Assuming an effect size of 0.15 (small effect size) across the 4 measurement moments (T0, T2, T4) between the two groups (group*time interaction), a total of 154 patients were needed, i.e. 77 per group. This was based on a Repeated measures ANOVA with an alpha of 0.05, a power of 0.80 and a nonsphericity correction of 1, calculated with G*Power 3.1.9.7. To account for a 10% dropout, 77 patients per group will be included.

A previous study on intensified walking during cardiac rehabilitation after acute myocardial infarction showed a KvL-H increase of 0.9 at the time of discharge (our study: T3) to intake cardiac rehabilitation (our study: T4) from 5.2 to 6.1 at the time of T5. A KvL-H increase of at least 0.15 points is expected in our T-REX Twente sternal precautions group (intervention group); a minimal clinical difference corresponding to a standarized response mean of 0.2.

For the second primary endpoint, the relative percentage of daytime (between 6:00 and 23:00) non-bedtime up to and including 4 days postoperatively on the ICU and nursing ward is examined. From previous research in a similar population, it was observed that a relative rate of lying in bed of 60% is measured on day 1 after discharge from ICU, with a decrease of 6.5% per day (p < 0.001). Assuming a reduction on day 1 to 50%, the medium f2 effect size of 0.5 with a linear mixed model, two-sided testing, alpha of 0.05, power of 0.80 and two predictors (time and group), results in 14 patients needed per group.

The highest number of patients will be retained, i.e. 77 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are preoperatively included if they are undergoing a total median sternotomy at Thorax Centrum Twente (TCT)
* Patients with their treating cardiologist also working for TCT.

Exclusion Criteria:

* >72 hours of admission to the Intensive Care Unit (ICU)
* Postoperative delirium (diagnosed with Diagnostic and Statistical Manual of Mental Disorders (DSM) version V
* Patients with dementia (or other significant cognitive disorders)
* Dutch language barriers
* Patients with a cardiologist from a location other than TCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life after Myocardial Infarction Questionnaire (MacNew QLMI) | Preoperative to start of cardiac rehabilitation (4-6 weeks postoperatively)
  The first primary endpoint is the standardized response mean difference of Quality of Life after Myocardial Infarction Questionnaire (MacNew QLMI) pre-operative until the start of cardiac rehabilitation (4-6 weeks postoperatively).
  MacNew QLMI scores on a 7-pointscale (1-7), where 1 = always and 7 = never. MacNew QLMI is an ordinal scale, with a total sumscore of 189 points as the maximum quality of life.
Not lying in bed | Postoperative day 0 to postoperative day 4
  The second primary endpoint is the duration of not being in bed for up to 4 days in the ICU and the general ward, measured using two AX3 accelerometers.

SECONDARY OUTCOMES:
Numeric (Pain) Rating Scale (NPRS) | Preoperative to end of cardiac rehabilitation (12 weeks postoperatively)
  Difference in experienced pain (self-reported) as measured with NPRS It is an 11-point ordinal scale (0-10) with 0 = no pain whatsoever, 10 = the worst pain most pain imaginable.
Quality of Life after Myocardial Infarction Questionnaire (MacNew QLMI) | Preoperative to end of cardiac rehabilitation (12 weeks postoperatively)
  Difference in QoL as measured with MacNew QLMI. MacNew QLMI scores on a 7-pointscale (1-7), where 1 = always and 7 = never. MacNew QLMI is an ordinal scale, with a total sumscore of 189 points as the maximum quality of life.
Tampa Scale for Kinesiophobia (TSK) | Preoperative to end of cardiac rehabilitation (12 weeks postoperatively)
  Difference in kinesiophobia as measured with TSK. The questionnaire consists of 17 items where a higher score represents a higher degree of fear of movement.
Individual mobilisation activities as measured with AX3 Accelerometer | Postoperative (directly after surgery, day 0) until hospital discharge (expected to be around postoperative day 5 to a maximum of 7 days)
  During clinical admission immediately postoperatively, two AX3 accelerometers are placed on the patient, one lateroproximal on the right upper arm and one anterodistal on the right upper leg.
  Mobilisation activities include: lying in bed, sitting on a chair, standing, walking, cycling on a bike ergometer, walking the stairs.
Composite endpoint of sternal refixation, superficial and deep sternal wounds for 30 days after surgery | 30-days postoperative
  Definitions according to Netherlands Heart Registration

CONTACTS AND LOCATIONS:
Overall Officials: Frank R. Halfwerk, MD, PhD, Principal Investigator — Medisch Spectrum Twente, Enschede, the Netherlands
Locations (1):
- Thoraxcentrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be a plan to make individual participant data (IPD) available.
  Study protocol and statistical analysis plan might be published.
Supporting Information: Study Protocol, SAP
Time Frame: Protocol is expected to be submitted for publication in 2024
Access Criteria: Principal Investigator generally supports Open Access publishing and data sharing.

REFERENCES:
- [Background] Benning MM, Kuo JM, Raushel FM, Holden HM. Three-dimensional structure of phosphotriesterase: an enzyme capable of detoxifying organophosphate nerve agents. Biochemistry. 1994 Dec 20;33(50):15001-7. doi: 10.1021/bi00254a008. PMID 7999757
- [Background] Floch HA. [Leprosy in Guadeloupe]. Bull Soc Pathol Exot Filiales. 1972 Jan-Feb;65(1):35-46. No abstract available. French. PMID 4677872
- [Background] Park L, Coltman C, Agren H, Colwell S, King-Shier KM. "In the tube" following sternotomy: A quasi-experimental study. Eur J Cardiovasc Nurs. 2021 Feb 1;20(2):160-166. doi: 10.1177/1474515120951981. PMID 33611341
- [Background] Holloway C, Pathare N, Huta J, Grady D, Landry A, Christie C, Pierce P, Bopp C. The Impact of a Less Restrictive Poststernotomy Activity Protocol Compared With Standard Sternal Precautions in Patients Following Cardiac Surgery. Phys Ther. 2020 Jul 19;100(7):1074-1083. doi: 10.1093/ptj/pzaa067. PMID 32302408